CLINICAL TRIAL: NCT00780208
Title: The Evaluation of the Safety and Efficacy of the Methylphenidate Patch in Former Stimulant Users With ADHD
Brief Title: Evaluating the Methylphenidate Patch to Treat Former Stimulant Users With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Aimee McRae-Clark, Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR#16784
Record Dates: First submitted 2008-10-23; First posted 2008-10-27 (Estimated); Results first posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Adult Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Attention Deficit Hyperactivity ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Daytrana (methylphenidate patch) (Other): Methylphenidate patch
  Interventions: Drug: Daytrana (methylphenidate patch)

INTERVENTIONS:
Drug: Daytrana (methylphenidate patch) — Subjects will be provided with a 7-day supply of medication at each study visit. The dose will be flexible and will be titrated based on effect and tolerability. Unless a subject is experiencing side effects, the dose will be increased if a 25% reduction in ADHD symptoms as determined by the WRAADDS is not obtained. A proposed dosing schedule is as follows: Week 1: 12.5 cm2, Week 2: 18.75 cm2, Week 3: 25 cm2, Week 4: 37.5 cm2. The dose may be decreased as needed for tolerability.
  Other Names: Daytrana Patch, Methylphenidate Patch

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of Daytrana® in the treatment of attention deficit hyperactivity disorder (ADHD) in adults who have abused stimulants in the past. Daytrana® is a stimulant medication that has been approved by the Food and Drug Administration for the treatment of ADHD in children over the age of 6 years old.

DETAILED DESCRIPTION:
Methylphenidate and amphetamines are considered to be the first line of treatment for ADHD in children (Biederman et al, 1997). Although treating children and adolescents with stimulants does not appear to increase the risk of substance use disorders (Wilens et al, 2003), little is known about the abuse of prescription stimulants in adults with ADHD. A review of the literature on the abuse potential of methylphenidate in animals and humans found that methylphenidate produced reinforcing, discriminative-stimulus, and subjective effects similar to amphetamines or cocaine (Kollins et al, 2001). Although the abuse rates of methylphenidate and other stimulant medications used for the treatment of ADHD have not been empirically established, significant concern exists so that regulatory mandates are enforced to control distribution, and some physicians may be reluctant to use stimulants in patients with drug abuse histories. The introduction of a methylphenidate patch is an important advancement, as the patch formulation should increase compliance while minimizing abuse potential, making it an attractive treatment option in the large population of individuals who have a history of previous drug misuse. The primary aim of this study is to assess the efficacy of the methylphenidate patch in adult individuals with ADHD who have abused stimulants in the past. It is hypothesized that the methylphenidate patch will be efficacious in reducing ADHD symptoms in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women, 18 to 65 years of age
2. Meet DSM-IV criteria for past stimulant (cocaine, methamphetamine, or prescription stimulant) abuse or dependence, with past abuse/dependence defined as a minimum of three months since meeting DSM-IV criteria, or have exhibited a pattern of stimulant misuse. For the purposes of this study, stimulant misuse will be defined as using someone else's stimulant ADHD medication for a minimum of four times in a one-month period, and this misuse must have occurred for at least three months.
3. Meet DSM-IV criteria for current ADHD, determined by a clinical interview and confirmed by semi-structured interview with the Conners' Adult ADHD Diagnostic Interview for DSM-IV (CAAR-D; Conners et al, 1999)
4. ADHD symptom severity indicated by a score of 12 or greater on the Wender-Reimherr Adult Attention Deficit Disorder Scale
5. All subjects will agree to and sign a written, IRB-approved informed consent
6. Subjects must live within a 60-mile radius of Charleston, SC, to facilitate study visit compliance

Exclusion Criteria:

1. Individuals meeting DSM-IV dependence for any substance with the exception of nicotine and caffeine
2. Individuals meeting DSM-IV criteria for a lifetime history of schizophrenia or another non-affective psychotic disorder or bipolar disorder, since these patients will most likely be taking other psychotropic medications and often require intensive psychiatric care
3. Individuals meeting DSM-IV criteria for current major depressive disorder or eating disorder, since these individuals will likely require treatment with psychotropic medications.
4. Individuals who present significant suicidal risk
5. Individuals with significant cognitive impairment as measured by a score of less than 26 on the Mini-Mental Status Exam, as they may be unable to understand the informed consent, comply with study protocol, or accurately complete assessments
6. Individuals currently receiving stimulants, benzodiazepines, antidepressant or antipsychotic medications.
7. Individuals currently receiving psychotherapy focusing on reducing ADHD symptoms, as this could confound the effects of methylphenidate treatment
8. Pregnant or nursing women, or women who refuse to use adequate birth control, as methylphenidate has not been approved for use in pregnancy
9. Individuals without stable housing, as contacting these individuals would be difficult
10. Individuals with major medical illnesses (e.g., HIV, renal failure, unstable angina, chronic obstructive pulmonary disease, infectious hepatitis)
11. Patients with uncontrolled hypertension (defined as having blood pressure greater than 140/90 measured on 3 or more occasions), as methylphenidate treatment can be associated with increases in blood pressure
12. Individuals with a significant family history of cardiac abnormalities, as these individuals may be more susceptible to cardiac adverse events
13. Individuals who are obese (greater than 30% over ideal weight or BMI greater than 30) as this may interfere with absorption of methylphenidate
14. Individuals who, in the investigators' opinion, would not be able to comply with study procedures, such as individuals unable to reliably present for intake appointments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-04; Primary Completion 2008-10 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee L. McRae-Clark, Pharm.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Daytrana (Methylphenidate Patch)
Started | 14
Completed | 8
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Daytrana (Methylphenidate Patch)
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 28.5 [22 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: ADHD Symptom Severity
Description: Primary efficacy endpoint will be ADHD symptom severity, as measured by mean change from baseline in the Wender-Reimherr Adult Attention Deficit Disorder Scale total score (WRAADS).The WRAADS measures symptoms in 7 categories: attention difficulties, hyperactivity/restlessness, temper, affective lability, emotional overreactivity, disorganization, and impulsivity. The scale rates individual items from 0 to 2 (0 = not present, 1 = mild, 2 = clearly present) so there may be a minimum total score of 0 (no symptoms present) through a maximum score of 56 (symptoms clearly present).
Time Frame: Baseline, Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daytrana (Methylphenidate Patch)
Number analyzed (Participants) | 14
units on a scale | -17.93 (5.89)

2. Secondary Outcome: Number of Participants With Positive Drug Screen
Description: Secondary efficacy endpoints will be substance use during the study, as measured by total number of participants testing positive for substances other than a stimulant on weekly urine drug screens
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Daytrana (Methylphenidate Patch)
Number analyzed (Participants) | 14
Participants | 4

ADVERSE EVENTS:
Arm/Group | Daytrana (Methylphenidate Patch)
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 10/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daytrana (Methylphenidate Patch) (N=14)
Skin reaction (Skin and subcutaneous tissue disorders) | 8 (9)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (General disorders) | 4 (5)
Sinus/cold/allergies (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry mouth (General disorders) | 2 (2)
Canker sores (Skin and subcutaneous tissue disorders) | 1 (1)
Paresthesia (General disorders) | 1 (2)
Insomnia (General disorders) | 1 (1)
Hyperactivity (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Yeast infection (Infections and infestations) | 1 (1)
Tooth pain (General disorders) | 1 (1)
Hot flash (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size and open-label design, preliminary nature of the trial precludes the ability to make treatment recommendations based on the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes